CLINICAL TRIAL: NCT05882357
Title: A Phase 3, Open-label Study Evaluating the Pharmacokinetics, Safety, and Tolerability of Elexacaftor/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects 12 to Less Than 24 Months of Age
Brief Title: Evaluation of Elexacaftor/Tezacaftor/Ivacaftor (ELX/TEZ/IVA) in Cystic Fibrosis (CF) Participants 12 to Less Than 24 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VX22-445-122; 2023-503230-49-00 (Other: EU CT)
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A (Experimental): Participants will receive ELX/TEZ/IVA in the morning and IVA in the evening.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA
- Part B (Experimental): Participants will receive ELX/TEZ/IVA in the morning and IVA in the evening with the dose(s) to be based on the outcome of Part A.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination granules for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Granules for oral administration
  Other Names: VX-770; ivacaftor

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, tolerability, pharmacodynamics (PD), and efficacy of ELX/TEZ/IVA in CF subjects 12 to less than (<) 24 months of age.

ELIGIBILITY:
Key Inclusion Criteria:

Participants who have at least 1 F508del mutation in the CF transmembrane conductance regulator (CFTR) gene or another ELX/TEZ/IVA-responsive CFTR mutation

Key Exclusion Criteria:

History of any illness or any clinical condition that, in the opinion of the investigator, might either confound the results of the study or pose an additional risk in administering study drug(s) to the participant

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Part A: Observed Pre-dose Concentration (Ctrough) of ELX, TEZ, IVA, and their Relevant Metabolites | Day 1 up to Day 15
Part A: Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 43
Part B: Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Week 28

SECONDARY OUTCOMES:
Part B: Observed Pre-dose Concentration (Ctrough) of ELX, TEZ, IVA, and their Relevant Metabolites | Day 15 up to Week 16
Part B: Absolute Change in Sweat Chloride (SwCl) | From Baseline Through Week 24

CONTACTS AND LOCATIONS:
Locations (19):
- Australia (4):
  - Telethon Kids Institute, Nedlands
  - The Royal Children's Hospital, Parkville
  - Queensland Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- Juliane Marie Center, Rigshospitalet, Copenhagen, Denmark
- Germany (3):
  - Charite Paediatric Pulmonology Department, Berlin
  - Kinderklinik III, Abt. fur Pneumologie, Essen
  - Medizinische Hochschule Hannover, Hanover
- Erasmus Medical Center / Sophia Children's Hospital, Rotterdam, Netherlands
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Kinderspital Zuerich, Zurich
- United Kingdom (6):
  - Children and Young Adults Research Unit, Cardiff
  - Leeds General Infirmary, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Children, London
  - Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing